CLINICAL TRIAL: NCT07087561
Title: The Effects and Mechanisms of Short-Term Nutritional Enhancement Combined With Health Education on Clinical Outcomes in Postoperative Patients With Colorectal Cancer: A Multicenter, Open-Label, Randomized Controlled Trial
Brief Title: Short-Term Nutritional Enhancement Combined With Health Education in Postoperative Colorectal Cancer Patients: A Randomized Controlled Trial
Acronym: NUTRI-CRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaoqin Luo (Other)
Responsible Party: Sponsor-Investigator, Xiaoqin Luo, Professor, Xi'an Jiaotong University
Organization: Xi'an Jiaotong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: No: XJTU1AF2025LSYY-016
Record Dates: First submitted 2025-07-18; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer (Diagnosis); Malnutrition or Risk of Malnutrition
Keywords: Colorectal Cancer; Nutrition Support; Health Education; Patient-Reported Outcomes; Nutritional Risk; Cancer Rehabilitation; Randomized Controlled Trial
MeSH Terms: conditions — Colorectal Neoplasms; Disease; Malnutrition; Health Education

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, open-label, parallel-group randomized controlled trial involving four intervention arms. Participants are assigned in a 1:1:1:1 ratio to one of the following: (A) short-term nutritional enhancement combined with health education, (B) health education alone, (C) nutritional enhancement alone, or (D) standard care. Stratified randomization is performed based on baseline nutritional status and cancer stage to ensure group balance.
Masking Description: Laboratory personnel conducting metabolomic, microbiome, and single-cell analyses will remain blinded to group allocation to reduce bias during data generation and interpretation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nutritional Enhancement Plus Health Education (Experimental): Participants in this arm will receive individualized nutritional enhancement along with structured health education. Nutritional intervention includes personalized dietary plans and oral nutritional supplements based on energy and protein requirements. Health education is delivered via an "Internet Plus" platform and includes weekly videos and interactive content focusing on nutrition, physical activity, and psychological support. The intervention lasts for 14 days and is followed by a 12-month, and annually up to 5 years to evaluate both clinical outcomes and biological markers of response. follow-up period.
  Interventions: Dietary Supplement: Personalized Oral Nutritional Supplementation; Drug: Personalized Parenteral Nutritional Supplementation; Behavioral: Structured Nutrition-Focused Health Education
- Health Education Only (Experimental): Participants in this arm will receive structured health education without additional nutritional supplementation. The education is delivered via an "Internet Plus" platform, including weekly videos and interactive content focused on nutrition knowledge, physical activity guidance, and psychological support. This intervention is administered for 14 days, followed by a 12-month follow-up and annually up to 5 years.
  Interventions: Behavioral: Structured Nutrition-Focused Health Education
- Nutritional Enhancement Only (Experimental): Participants in this arm will receive individualized nutritional enhancement based on personalized dietary assessment and calculated energy and protein needs. Interventions include oral nutritional supplements and tailored dietary counseling provided by a clinical nutrition team. No additional health education is provided. The intervention phase lasts for 14 days, with scheduled follow-up for 12 months and annually up to 5 years.
  Interventions: Dietary Supplement: Personalized Oral Nutritional Supplementation; Drug: Personalized Parenteral Nutritional Supplementation
- Standard Care (Control) (No Intervention): Participants in this arm will receive standard inpatient care without structured nutritional intervention or health education. Patients eat according to personal ability and appetite but do not receive individualized nutrition counseling or supplemental nutrition support. This group serves as the control group for comparison. Routine clinical follow-up will be conducted for 12 months and annually up to 5 years.

INTERVENTIONS:
Dietary Supplement: Personalized Oral Nutritional Supplementation — Participants receive individualized oral nutritional supplementation based on energy and protein requirements, calculated using the Harris-Benedict equation and body weight (1.2-1.5 g protein/kg/day). The supplement may include complete nutrition powder, whey protein powder, and compound multivitamins. The intervention is prescribed and monitored by a clinical nutrition team and adjusted every 3 days during the 14-day intervention phase. The goal is to ensure both energy and protein intake targets are met. Supplements are administered in addition to standard meals.
  Other Names: ONS
  Arms: Nutritional Enhancement Only; Nutritional Enhancement Plus Health Education
Drug: Personalized Parenteral Nutritional Supplementation — For participants unable to meet nutritional goals through oral intake, parenteral nutrition is administered intravenously. The formulation includes amino acids, glucose, lipids, electrolytes, trace elements, and vitamins. Dosages are aligned with those of the enteral nutrition group, ensuring a consistent intake of energy and protein (1.2-1.5 g/kg/day protein). Formulation and administration follow standardized hospital protocols and are supervised by the nutrition support team.
  Other Names: PN
  Arms: Nutritional Enhancement Only; Nutritional Enhancement Plus Health Education
Behavioral: Structured Nutrition-Focused Health Education — Participants receive structured health education focused on nutrition, physical activity, and psychological well-being. The education is delivered over 14 days using a digital "Internet Plus" platform, featuring weekly videos, interactive Q&A sessions, and guidance from a multidisciplinary nutrition support team. Educational content covers dietary recommendations, exercise safety, stress management, and post-treatment recovery strategies. Materials are updated weekly, and participants may access them remotely via smartphone or tablet. This intervention aims to improve nutrition knowledge, adherence, and health behavior change.
  Other Names: Internet-Based Health Education; Multimedia Health Literacy Intervention
  Arms: Health Education Only; Nutritional Enhancement Plus Health Education

SUMMARY:
This clinical study aims to evaluate whether short-term personalized nutritional support, when combined with structured health education, can improve nutritional status, quality of life, and clinical outcomes in patients who have undergone surgery for colorectal cancer (CRC). Colorectal cancer is one of the most common cancers worldwide, and many patients experience malnutrition and poor physical condition during treatment, which can negatively affect recovery and long-term survival.

In this multicenter, randomized, controlled clinical trial, approximately 360 postoperative CRC patients will be enrolled and randomly assigned to one of four groups: (A) nutritional enhancement combined with health education, (B) health education alone, (C) nutritional enhancement alone, or (D) standard care (control group). Nutritional support will include individualized diet counseling and oral nutritional supplements tailored to each patient's needs. Health education will be delivered using an "Internet Plus" approach, including weekly educational videos and expert consultations focusing on nutrition, physical activity, and mental health.

The primary objectives are to determine whether these interventions can improve patients' short-term nutritional status and quality of life. Secondary outcomes include the impact of interventions on long-term survival, treatment-related side effects, patient adherence to nutrition recommendations, and psychological well-being.

This study will also investigate the biological mechanisms underlying the clinical effects by analyzing changes in the gut microbiome, blood-based metabolic profiles, and immune responses. Blood, stool, and tumor tissue samples will be collected and analyzed using advanced techniques, including untargeted metabolomics, metagenomics, and single-cell sequencing.

This trial is designed to provide evidence for the integration of nutritional strategies into routine cancer care, and to guide the development of more personalized, effective nutrition-based therapies for colorectal cancer patients. Participants will be followed for up to annually up to 5 years to evaluate both clinical outcomes and biological markers of response.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, randomized controlled clinical trial designed to assess the effects and underlying mechanisms of short-term nutritional enhancement combined with health education on clinical outcomes in patients undergoing surgery for non-metastatic colorectal cancer (stages IIa, IIb, IIIa). The rationale is based on the high prevalence of malnutrition among CRC patients, which significantly impacts treatment tolerance, quality of life, and long-term prognosis.

Eligible participants will be randomized into four parallel arms: (1) individualized nutritional enhancement plus structured health education; (2) structured health education alone; (3) individualized nutritional enhancement alone; and (4) standard care without additional intervention. Personalized nutrition plans will be developed based on energy and protein needs, supported by dietary counseling and the provision of oral nutritional supplements. Health education will be delivered through a digital platform, featuring weekly videos and interactive content on nutrition, exercise, and psychological well-being.

The study includes a 14-day intervention phase and a 12-month follow-up period. Outcomes will be assessed at baseline, and at 1, 2, 3, 6, and 12 months, and annually up to 5 years to evaluate both clinical outcomes and biological markers of response.post-intervention. Key endpoints include improvements in nutritional status, patient-reported quality of life, and overall survival metrics.

To investigate mechanisms, the study incorporates biological sampling and multi-omics analysis. Non-targeted serum metabolomics, gut microbiota metagenomics, and single-cell RNA sequencing of tumor and adjacent normal tissues will be used to characterize metabolic and immune changes associated with the interventions. The study also evaluates the role of inflammatory markers and immune cell profiles in mediating clinical effects.

This trial is expected to generate high-quality evidence supporting the integration of nutrition and health education strategies into standard postoperative care for CRC patients. It may also identify novel metabolic or microbial biomarkers associated with treatment response and prognosis, contributing to the development of precision nutrition approaches in oncology.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* Pathologically confirmed diagnosis of colon or rectal cancer
* Mentally alert and capable of communication
* Willing to participate in follow-up, with an estimated life expectancy of more than 6 months
* Cancer stage IIa, IIb, or IIIa

Exclusion Criteria:

* Nutritional risk screening score of mPG-SGA < 2 or NRS-2002 < 3
* Diagnosed with AIDS
* History of organ transplantation
* Pregnant or breastfeeding women
* Concurrent participation in another interventional clinical trial
* Inability to care for oneself independently
* Inability to engage in physical activity during the perioperative period
* Severe comorbid conditions (e.g., uncontrolled cardiovascular disease, severe hepatic or renal dysfunction)
* Known allergy or intolerance to components of the nutritional supplements used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2029-10-10 (Estimated); Study Completion 2030-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in Nutritional Status Assessed by Modified Patient-Generated Subjective Global Assessment (mPG-SGA) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Longitudinal assessment of nutritional status using the mPG-SGA, a validated tool composed of five sections (weight loss history, dietary intake, symptoms, function/activity, and age). Total scores range from 0 to ≥7 points, with higher scores indicating worse nutritional status. Patients will be classified as:
  0-2 = Normal
  3-6 = Mild malnutrition
  ≥7 = Moderate to severe malnutrition.
Change in Global Health Status Score on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Assessment of patients' perceived overall health status using the global health subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Scores range from 0 to 100, with higher scores indicating better global quality of life.
Change in Symptom Scores on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Assessment of symptom burden including fatigue, pain, nausea/vomiting, appetite loss, sleep disturbance, constipation, diarrhea, and financial difficulty using symptom subscales of the EORTC QLQ-C30. Each symptom is scored separately from 0 to 100, with higher scores indicating worse symptom severity.
Overall Survival (OS) in Cancer Patients | From date of enrollment until death or last follow-up (up to 5 years)
  Overall survival is defined as the time from the date of enrollment to the date of death from any cause. Patients still alive at the last follow-up will be censored. Kaplan-Meier survival analysis and Cox proportional hazards regression will be used to estimate survival and explore associations with baseline and longitudinal nutritional status.
Progression-Free Survival (PFS) in Cancer Patients | From date of enrollment until death or last follow-up (up to 5 years)
  Progression-free survival is defined as the time from enrollment to the first documented disease progression or death from any cause, whichever occurs first. Patients without progression at the time of last follow-up will be censored. PFS will be analyzed using Kaplan-Meier estimates and Cox regression models, stratified by nutritional status.

SECONDARY OUTCOMES:
Change in Nutritional Risk Assessed by Nutritional Risk Screening 2002 (NRS-2002) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Longitudinal evaluation of nutritional risk using the NRS-2002, which considers disease severity, nutritional impairment, and age. Total score ranges from 0 to ≥7 points. A score of ≥3 indicates nutritional risk and warrants intervention; <3 indicates no immediate risk.
Serum Total Protein | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Serum total protein concentration (g/L), used to evaluate protein-energy nutritional status. Measured using standard biochemical assays.
Serum Albumin | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Serum albumin concentration (g/L), used to assess visceral protein status and systemic inflammation.
Serum Prealbumin | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Serum prealbumin level (mg/L), an indicator of short-term changes in protein-energy nutritional status.
Serum Transferrin | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Serum transferrin concentration (g/L), a marker of protein status and iron metabolism.
C-Reactive Protein (CRP) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Serum CRP (mg/L), a marker of systemic inflammation and acute-phase response.
Blood Glucose | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Fasting blood glucose (mmol/L), measured to assess metabolic function and risk of hyperglycemia.
Aspartate Aminotransferase (AST) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  AST concentration (U/L), used as a liver function test and hepatotoxicity marker.
Alanine Aminotransferase (ALT) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  ALT level (U/L), a liver enzyme measured to monitor hepatic injury.
Interleukin-1 (IL-1) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  IL-1 concentration (pg/mL), a pro-inflammatory cytokine indicative of immune and inflammatory activity.
Tumor Necrosis Factor-alpha (TNF-α) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Tumor Necrosis Factor-alpha (TNF-α) level (pg/mL) measured to assess systemic inflammation and cancer-related cachexia.
Serum Creatinine | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Serum creatinine (μmol/L), measured to evaluate kidney function and treatment-related nephrotoxicity.
Blood Urea Nitrogen | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Blood urea nitrogen (umol/L), used to monitor renal function and protein catabolism.
Total Bilirubin | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Blood urea nitrogen (umol/L), used to monitor renal function and protein catabolism.
Total Cholesterol | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Total cholesterol level (mmol/L), measured to assess lipid metabolism and nutritional status.
Triglycerides | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Serum triglyceride level (mmol/L), used to evaluate energy reserves and lipid metabolism.
High-Density Lipoprotein Cholesterol (HDL-C) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  HDL-C (mmol/L), assessed as a marker of cardiovascular health and lipid status.
Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  LDL-C (mmol/L), measured as a risk factor for cardiovascular disease and lipid status.
Interleukin-6 (IL-6) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  IL-6 level (pg/mL), a pro-inflammatory cytokine measured to monitor systemic inflammation and cachexia.
Hemoglobin | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Hemoglobin concentration (*10⁹/L), used to assess anemia and oxygen-carrying capacity.
White Blood Cell Count (Leukocytes) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Total white blood cell count (*10⁹/L), measured to monitor immune status and detect infection or myelosuppression.
Neutrophil Count | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Absolute neutrophil count (*10⁹/L), used to assess infection risk and bone marrow suppression.
Lymphocyte Count | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Lymphocyte count (*10⁹/L), measured to evaluate immune competence.
Red Blood Cell Count | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Red blood cell count (*10¹²/L), used to assess erythropoiesis and anemia.
Platelet Count | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Platelet count (*10⁹/L), measured to evaluate coagulation status and myelosuppression.
Height | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Standing height (cm) measured using a stadiometer with 0.5 cm precision. Values adjusted for presence of ascites, edema, or large tumors.ascites, systemic edema, and huge tumors.
Body Weight | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Body weight (kg) measured using a calibrated scale with 0.2 kg precision. Values adjusted if ascites or edema are present.
Body Mass Index (BMI) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  BMI calculated as weight (kg) divided by height squared (m²), recorded to one decimal place.
Change in Anxiety Symptoms Assessed by Hospital Anxiety and Depression Scale (HADS-A) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Assessment of anxiety using the HADS-A subscale of the Hospital Anxiety and Depression Scale. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms. Results will be analyzed in relation to nutritional status (normal, mild, moderate malnutrition).
Change in Depression Symptoms Assessed by Hospital Anxiety and Depression Scale (HADS-D) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Assessment of depressive symptoms using the HADS-D subscale of the Hospital Anxiety and Depression Scale. Scores range from 0 to 21, with higher scores indicating more severe depression. Results will be analyzed in relation to nutritional status (normal, mild, moderate malnutrition).
Functional Performance Measured by Karnofsky Performance Status (KPS) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Functional performance will be evaluated using the Karnofsky Performance Status (KPS) scale, which ranges from 0 to 100. Higher scores indicate better functional ability and independence in daily activities. Longitudinal KPS changes will be assessed in relation to changes in nutritional status over time.
Changes in Sleep Quality Assessed by Pittsburgh Sleep Quality Index (PSQI) | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Sleep quality and disturbances will be evaluated using the Pittsburgh Sleep Quality Index (PSQI), a standardized questionnaire assessing seven components of sleep. Total scores range from 0 to 21, with higher scores indicating poorer sleep quality. PSQI scores will be analyzed in relation to nutritional risk categories and treatment phases.
Changes in Physical Activity Level During Cancer Treatment | Baseline, after the intervention, 1, 2, 3, 6, and 12 months after intervention; annually up to 5 years
  Assessment of leisure-time physical activity levels (mild, moderate, vigorous) and their relationship with nutritional status and cancer treatment response.
Changes in Nutrition-Related Knowledge, Attitudes, and Practices (KAP) | Baseline, after the intervention, 6 months after intervention; annually up to 5 years
  Patients' dietary knowledge, attitudes, and practices will be assessed using a validated Nutrition KAP (Knowledge, Attitude, and Practice) questionnaire. The total score ranges from 0 to 104, with higher scores indicating better nutritional knowledge, more positive attitudes, and healthier dietary behaviors. Longitudinal changes in KAP scores will be evaluated in relation to treatment outcomes.
Healthcare Utilization and Cost of Nutrition-Related Care | From admission through 30-day post-discharge and annually for 5 years
  Evaluation of healthcare utilization related to nutritional care, including total number of hospitalization days, number of ICU admissions, and direct costs associated with enteral and parenteral nutrition support. Metrics will be analyzed in relation to malnutrition risk at baseline and during treatment.
Incidence of Serious Adverse Events Related to Nutrition or Treatment | Continuously from enrollment through end of study follow-up (up to 5 years)
  Tracking of serious adverse events potentially related to nutritional support or treatment, including infections, allergic reactions, gastrointestinal distress, and metabolic complications.

OTHER OUTCOMES:
Predictive Value of Baseline Nutritional Indicators for 30-Day Clinical Events | Baseline to 30 days post-admission
  Evaluation of whether baseline nutritional indicators-including mPG-SGA scores and laboratory biomarkers such as albumin, prealbumin, and CRP-predict 30-day clinical outcomes, including mortality, ICU admission, and significant unintentional weight loss (>5%). Logistic regression will be used for model construction and discrimination.
Nutritional Trajectory Typing and Clustering | From baseline to 12-month follow-up
  Identification of distinct nutritional change trajectories over time using latent class growth analysis (LCGA) and hierarchical clustering based on serial measurements of mPG-SGA and anthropometric data. Trajectories will be used to classify patients into nutritional risk subgroups.
Agreement Between Nutritional Screening Tools (mPG-SGA vs. NRS-2002) | Baseline and each scheduled follow-up (up to 5 years)
  Assessment of the diagnostic agreement, sensitivity, and specificity of two nutritional screening tools-modified Patient-Generated Subjective Global Assessment (mPG-SGA) and Nutritional Risk Screening 2002 (NRS-2002)-in detecting malnutrition risk. Agreement will be evaluated using Cohen's kappa and ROC curve analysis.
Sociodemographic Determinants of Malnutrition | From baseline throughout study follow-up (up to 5 years)
  Analysis of sociodemographic factors-including income level, education, employment status, and rural vs. urban residence-in predicting baseline malnutrition and nutritional deterioration over time. Multivariable models will be used to explore independent associations.
Patient Adherence to Out-of-Hospital Nutritional Support | Baseline to 12 months post-treatment initiation
  Evaluation of patient-reported adherence to prescribed oral nutritional supplements or enteral/parenteral support regimens after hospital discharge. Adherence data will be collected via structured interviews and compared with clinical outcomes and readmission rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Xi 'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The study intends to share IPD with other researchers for advancing scientific understanding and improving patient care. The shared data will include anonymized participant information, such as demographic details, clinical outcomes, and treatment responses. The data will be stripped of any identifiers to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available after the publication of the main study results, anticipated to be by the end of 2030. The data will be accessible for a period of five years following this date.
Access Criteria: Researchers interested in accessing the data will be required to submit a proposal outlining their intended use of the data, which will be reviewed by the study's principal investigator. Access will be granted based on the scientific merit and ethical considerations of the proposal.

REFERENCES:
- [Background] Yang Y, Han Z, Li X, Huang A, Shi J, Gu J. Epidemiology and risk factors of colorectal cancer in China. Chin J Cancer Res. 2020 Dec 31;32(6):729-741. doi: 10.21147/j.issn.1000-9604.2020.06.06. PMID 33446996
- [Background] Bennell KL, Lawford BJ, Keating C, Brown C, Kasza J, Mackenzie D, Metcalf B, Kimp AJ, Egerton T, Spiers L, Proietto J, Sumithran P, Harris A, Quicke JG, Hinman RS. Comparing Video-Based, Telehealth-Delivered Exercise and Weight Loss Programs With Online Education on Outcomes of Knee Osteoarthritis : A Randomized Trial. Ann Intern Med. 2022 Feb;175(2):198-209. doi: 10.7326/M21-2388. Epub 2021 Nov 30. PMID 34843383
- [Background] Ratri DMN, Hamidah KF, Puspitasari AD, Farid M. Video-based health education to support insulin therapy in diabetes mellitus patients. J Public Health Res. 2020 Jul 3;9(2):1849. doi: 10.4081/jphr.2020.1849. eCollection 2020 Jul 3. PMID 32728588
- [Background] Adam M, Young-Wolff KC, Konar E, Winkleby M. Massive open online nutrition and cooking course for improved eating behaviors and meal composition. Int J Behav Nutr Phys Act. 2015 Dec 3;12:143. doi: 10.1186/s12966-015-0305-2. PMID 26630879
- [Background] Wang Y, Wang Y, Xu C, Liu Y, Huang Z. Identification of Novel Tumor-Microenvironment-Regulating Factor That Facilitates Tumor Immune Infiltration in Colon Cancer. Mol Ther Nucleic Acids. 2020 Aug 29;22:236-250. doi: 10.1016/j.omtn.2020.08.029. eCollection 2020 Dec 4. PMID 33230430
- [Background] Brown TE, Banks MD, Hughes BGM, Lin CY, Kenny LM, Bauer JD. Randomised controlled trial of early prophylactic feeding vs standard care in patients with head and neck cancer. Br J Cancer. 2017 Jun 27;117(1):15-24. doi: 10.1038/bjc.2017.138. Epub 2017 May 23. PMID 28535154
- [Background] Murphy JL, Munir F, Davey F, Miller L, Cutress R, White R, Lloyd M, Roe J, Granger C, Burden S, Turner L. The provision of nutritional advice and care for cancer patients: a UK national survey of healthcare professionals. Support Care Cancer. 2021 May;29(5):2435-2442. doi: 10.1007/s00520-020-05736-y. Epub 2020 Sep 12. PMID 32918612
- [Background] Liu Y, Zhang H, Dove WF, Wang Z, Zhu Z, Pickhardt PJ, Reichelderfer M, Li L. Quantification of Serum Metabolites in Early Colorectal Adenomas Using Isobaric Labeling Mass Spectrometry. J Proteome Res. 2023 May 5;22(5):1483-1491. doi: 10.1021/acs.jproteome.3c00006. Epub 2023 Apr 4. PMID 37014956
- [Background] Liu Y, Lau HC, Yu J. Microbial metabolites in colorectal tumorigenesis and cancer therapy. Gut Microbes. 2023 Jan-Dec;15(1):2203968. doi: 10.1080/19490976.2023.2203968. PMID 37095682
- [Background] Niekamp P, Kim CH. Microbial Metabolite Dysbiosis and Colorectal Cancer. Gut Liver. 2023 Mar 15;17(2):190-203. doi: 10.5009/gnl220260. Epub 2023 Jan 12. PMID 36632785
- [Background] Louis P, Hold GL, Flint HJ. The gut microbiota, bacterial metabolites and colorectal cancer. Nat Rev Microbiol. 2014 Oct;12(10):661-72. doi: 10.1038/nrmicro3344. Epub 2014 Sep 8. PMID 25198138
- [Background] Liu H, Lei W, Li Z, Wang X, Zhou L. NR3C2 inhibits the proliferation of colorectal cancer via regulating glucose metabolism and phosphorylating AMPK. J Cell Mol Med. 2023 Apr;27(8):1069-1082. doi: 10.1111/jcmm.17706. Epub 2023 Mar 23. PMID 36950803
- [Background] Tabata S, Kojima Y, Sakamoto T, Igarashi K, Umetsu K, Ishikawa T, Hirayama A, Kajino-Sakamoto R, Sakamoto N, Yasumoto KI, Okano K, Suzuki Y, Yachida S, Aoki M, Soga T. L-2hydroxyglutaric acid rewires amino acid metabolism in colorectal cancer via the mTOR-ATF4 axis. Oncogene. 2023 Apr;42(16):1294-1307. doi: 10.1038/s41388-023-02632-7. Epub 2023 Mar 6. PMID 36879117
- [Background] Ravasco P, Monteiro-Grillo I, Vidal PM, Camilo ME. Dietary counseling improves patient outcomes: a prospective, randomized, controlled trial in colorectal cancer patients undergoing radiotherapy. J Clin Oncol. 2005 Mar 1;23(7):1431-8. doi: 10.1200/JCO.2005.02.054. Epub 2005 Jan 31. PMID 15684319
- [Background] Lu Z, Fang Y, Liu C, Zhang X, Xin X, He Y, Cao Y, Jiao X, Sun T, Pang Y, Wang Y, Zhou J, Qi C, Gong J, Wang X, Li J, Tang L, Shen L. Early Interdisciplinary Supportive Care in Patients With Previously Untreated Metastatic Esophagogastric Cancer: A Phase III Randomized Controlled Trial. J Clin Oncol. 2021 Mar 1;39(7):748-756. doi: 10.1200/JCO.20.01254. Epub 2021 Jan 8. PMID 33417481
- [Background] Prabhu Das I, Baker M, Altice C, Castro KM, Brandys B, Mitchell SA. Outcomes of multidisciplinary treatment planning in US cancer care settings. Cancer. 2018 Sep 15;124(18):3656-3667. doi: 10.1002/cncr.31394. Epub 2018 Sep 14. PMID 30216477
- [Background] Ye J, Hu Y, Chen X, Chang C, Li K. Comparative Effects of Different Nutritional Supplements on Inflammation, Nutritional Status, and Clinical Outcomes in Colorectal Cancer Patients: A Systematic Review and Network Meta-Analysis. Nutrients. 2023 Jun 16;15(12):2772. doi: 10.3390/nu15122772. PMID 37375676
- [Background] Chang YT, Chen CC, Chang SC, Chang YY, Lin BW, Chen HH, Hsieh YY, Hsu HC, Hsieh MC, Kuan FC, Wu CC, Lu WC, Su YL, Liang YH, Chen JB, Huang SY, Huang CW, Wang JY. Efficacy and Safety of a Parenteral Nutrition Program for Patients with RAS Wild-Type Metastatic Colorectal Cancer Administered First-Line Cetuximab Plus Chemotherapy: A Propensity Score Matching Study. Nutrients. 2023 Jun 30;15(13):2971. doi: 10.3390/nu15132971. PMID 37447297
- [Background] Sequential Enteral and Parenteral Nutrition Support Assisted by Nutritional Risk Screening Improves Outcome in the Colorectal Cancer Patients Undergoing Radical Surgery
- [Background] Matthews CE, Moore SC, Arem H, Cook MB, Trabert B, Hakansson N, Larsson SC, Wolk A, Gapstur SM, Lynch BM, Milne RL, Freedman ND, Huang WY, Berrington de Gonzalez A, Kitahara CM, Linet MS, Shiroma EJ, Sandin S, Patel AV, Lee IM. Amount and Intensity of Leisure-Time Physical Activity and Lower Cancer Risk. J Clin Oncol. 2020 Mar 1;38(7):686-697. doi: 10.1200/JCO.19.02407. Epub 2019 Dec 26. PMID 31877085
- [Background] Zietarska M, Krawczyk-Lipiec J, Kraj L, Zaucha R, Malgorzewicz S. Chemotherapy-Related Toxicity, Nutritional Status and Quality of Life in Precachectic Oncologic Patients with, or without, High Protein Nutritional Support. A Prospective, Randomized Study. Nutrients. 2017 Oct 11;9(10):1108. doi: 10.3390/nu9101108. PMID 29019951
- [Background] Tan S, Meng Q, Jiang Y, Zhuang Q, Xi Q, Xu J, Zhao J, Sui X, Wu G. Impact of oral nutritional supplements in post-discharge patients at nutritional risk following colorectal cancer surgery: A randomised clinical trial. Clin Nutr. 2021 Jan;40(1):47-53. doi: 10.1016/j.clnu.2020.05.038. Epub 2020 Jun 2. PMID 32563599
- [Background] Muscaritoli M, Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Oldervoll L, Ravasco P, Solheim TS, Strasser F, de van der Schueren M, Preiser JC, Bischoff SC. ESPEN practical guideline: Clinical Nutrition in cancer. Clin Nutr. 2021 May;40(5):2898-2913. doi: 10.1016/j.clnu.2021.02.005. Epub 2021 Mar 15. PMID 33946039
- [Background] Cong MH, Li SL, Cheng GW, Liu JY, Song CX, Deng YB, Shang WH, Yang D, Liu XH, Liu WW, Lu SY, Yu L. An Interdisciplinary Nutrition Support Team Improves Clinical and Hospitalized Outcomes of Esophageal Cancer Patients with Concurrent Chemoradiotherapy. Chin Med J (Engl). 2015 Nov 20;128(22):3003-7. doi: 10.4103/0366-6999.168963. PMID 26608978
- [Background] Muscaritoli M, Corsaro E, Molfino A. Awareness of Cancer-Related Malnutrition and Its Management: Analysis of the Results From a Survey Conducted Among Medical Oncologists. Front Oncol. 2021 May 13;11:682999. doi: 10.3389/fonc.2021.682999. eCollection 2021. PMID 34055649
- [Background] Baracos VE. Cancer-associated malnutrition. Eur J Clin Nutr. 2018 Sep;72(9):1255-1259. doi: 10.1038/s41430-018-0245-4. Epub 2018 Sep 5. No abstract available. PMID 30185853
- [Background] Planas M, Alvarez-Hernandez J, Leon-Sanz M, Celaya-Perez S, Araujo K, Garcia de Lorenzo A; PREDyCES(R) researchers. Prevalence of hospital malnutrition in cancer patients: a sub-analysis of the PREDyCES(R) study. Support Care Cancer. 2016 Jan;24(1):429-435. doi: 10.1007/s00520-015-2813-7. Epub 2015 Jun 23. PMID 26099900
- [Background] Gellrich NC, Handschel J, Holtmann H, Kruskemper G. Oral cancer malnutrition impacts weight and quality of life. Nutrients. 2015 Mar 27;7(4):2145-60. doi: 10.3390/nu7042145. PMID 25825828
- [Background] Seo SH, Kim SE, Kang YK, Ryoo BY, Ryu MH, Jeong JH, Kang SS, Yang M, Lee JE, Sung MK. Association of nutritional status-related indices and chemotherapy-induced adverse events in gastric cancer patients. BMC Cancer. 2016 Nov 18;16(1):900. doi: 10.1186/s12885-016-2934-5. PMID 27863481
- [Background] Aaldriks AA, van der Geest LG, Giltay EJ, le Cessie S, Portielje JE, Tanis BC, Nortier JW, Maartense E. Frailty and malnutrition predictive of mortality risk in older patients with advanced colorectal cancer receiving chemotherapy. J Geriatr Oncol. 2013 Jul;4(3):218-26. doi: 10.1016/j.jgo.2013.04.001. Epub 2013 Apr 30. PMID 24070460
- [Background] Nutritional status and risk factors for malnutrition in CRC patients undergoing neoadjuvant therapy
- [Background] Hebuterne X, Lemarie E, Michallet M, de Montreuil CB, Schneider SM, Goldwasser F. Prevalence of malnutrition and current use of nutrition support in patients with cancer. JPEN J Parenter Enteral Nutr. 2014 Feb;38(2):196-204. doi: 10.1177/0148607113502674. PMID 24748626
- [Background] Argiles JM. Cancer-associated malnutrition. Eur J Oncol Nurs. 2005;9 Suppl 2:S39-50. doi: 10.1016/j.ejon.2005.09.006. PMID 16437757
- [Background] Han B, Zheng R, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2022. J Natl Cancer Cent. 2024 Feb 2;4(1):47-53. doi: 10.1016/j.jncc.2024.01.006. eCollection 2024 Mar. PMID 39036382
- [Background] Zhou J, Zheng R, Zhang S, Zeng H, Wang S, Chen R, Sun K, Li M, Gu J, Zhuang G, Wei W. Colorectal cancer burden and trends: Comparison between China and major burden countries in the world. Chin J Cancer Res. 2021 Feb 28;33(1):1-10. doi: 10.21147/j.issn.1000-9604.2021.01.01. PMID 33707923
- [Background] The epidemiology of colorectal cancer in China
- [Background] Morgan E, Arnold M, Gini A, Lorenzoni V, Cabasag CJ, Laversanne M, Vignat J, Ferlay J, Murphy N, Bray F. Global burden of colorectal cancer in 2020 and 2040: incidence and mortality estimates from GLOBOCAN. Gut. 2023 Feb;72(2):338-344. doi: 10.1136/gutjnl-2022-327736. Epub 2022 Sep 8. PMID 36604116
- [Background] Zheng R, Zhang S, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2016. J Natl Cancer Cent. 2022 Feb 27;2(1):1-9. doi: 10.1016/j.jncc.2022.02.002. eCollection 2022 Mar. PMID 39035212
- [Background] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- See also: World Health Organization. Cancer[EB/OL]. Cancer[2023-05-12]. — https://www.who.int/news-room/fact-sheets/detail/cancer
- See also: World Health Organization. Colorectal Cancer Awareness Month 2022 — https://www.iarc.who.int/featured-news/colorectal-cancer-awareness-month-2022/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT07087561/Prot_SAP_000.pdf